CLINICAL TRIAL: NCT00779701
Title: Strict Glycemic Control by Insulin Infusion:Observations on Emergency Department Initiation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TU10526
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Hyperglycemia
Keywords: Hyperglycemia; Glycemic control
MeSH Terms: conditions — Hyperglycemia | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): All subjects placed on insulin infusion.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin infusion titrated to patients blood glucose to maintain blood glucose between 80-110mg/dL

SUMMARY:
Glycemic control can be safely achieved in surgical and medical intensive care unit settings and has been shown to improve short and long-term clinical outcomes. As such, insulin infusion protocols are routinely used in the ICU setting. The investigators plan to establish the use of strict glycemic control in a heterogenous group of acutely ill patients in the ED setting. The investigators propose to study the aspects of implementing a strict glycemic control protocol in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Patients with blood glucose ≥130 mg% considered to be critically ill as defined by:

APACHE II score ≥9 (See Appendix 1) OR >2 SIRS criteria with lactate ≥ 4 or BP < 90mmHg despite one liter of fluid OR Evidence of Organ Dysfunction (see Appendix 1)

Exclusion Criteria:

* Patients requiring urgent interventional procedure (e.g. cardiac catheterization, dialysis) or surgery performed outside of the ED.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina T Gentile, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Infusion: All subjects placed on insulin infusion.
  Insulin: Insulin infusion titrated to patients blood glucose to maintain blood glucose between 80-110mg/dL
Period: Overall Study
Arm/Group | Insulin Infusion
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Insulin Infusion
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Glycemic Control
Time Frame: Study duration 6 hours. Blood glucose checked at 30 minutes then every 15 minutes until within target blood glucose range then every hour.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Insulin Infusion
Number analyzed (Participants) | 27
Minutes | 225 (48.8)

ADVERSE EVENTS:
Arm/Group | Insulin Infusion
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes